CLINICAL TRIAL: NCT03260062
Title: Pilot Intervention to Improve Language in Deaf Children With Cochlear Implants
Brief Title: Parent-Child Early Approaches to Raising Language Skills (PEARLS) Intervention
Acronym: PEARLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Ivette Cejas, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20150457; R21DC016265 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Deafness, Bilateral
Keywords: cochlear implants; language development; parenting intervention; maternal sensitivity; facilitative language techniques
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEARLS (Experimental): Participants in this arm will receive 10 1-hour weekly sessions of the PEARLS intervention
  Interventions: Behavioral: Parent-Child Early Approaches to Raising Language Skills
- Control (Active Comparator): Participants in this arm will receive 10 1-hour weekly sessions of the standard of care LSL Speech Therapy
  Interventions: Other: Standard Care Speech therapy

INTERVENTIONS:
Behavioral: Parent-Child Early Approaches to Raising Language Skills — The PEARLS intervention will teach parents evidence-based language strategies and sensitive parenting (e.g., warmth, respect for autonomy, linguistic stimulation) to promote language development in young deaf children with cochlear implants (CI).
  Arms: PEARLS
Other: Standard Care Speech therapy — Families will participate in auditory-verbal therapy, which is the standard speech therapy with children with hearing loss.
  Arms: Control

SUMMARY:
The purpose of this research study is to develop and evaluate a parent training program, which aims to improve language. The study is being conducted to see if teaching parents positive parenting techniques and behavior strategies will improve the rate of language development in children with cochlear implants when compared to standard speech therapy (e.g., auditory-verbal therapy).

ELIGIBILITY:
Inclusion Criteria:

1. children who are severely to profoundly deaf and a cochlear implant candidate,
2. children who are 12 to 48 months,
3. English or Spanish as primary language spoken at home,
4. families educating their children in spoken language,
5. children who pass the cognitive screening, scoring 75 or above on the screening measure

Exclusion Criteria:

1. parents who do not consent to being videotaped,
2. children with moderate to severe developmental delays (as assessed using the Battelle Developmental Inventory (BDI-2) 2nd Edition for children ages 0 to 24 months or the Leiter International Performance Scale-Revised),
3. children with significant syndromes (e.g., CHARGE, autism, cerebral palsy) or severe brain abnormalities,
4. families who do not receive their auditory-verbal therapy from University of Miami (UM). Further, children who have already completed the BDI-2 within the past year as part of their Early Steps (Florida Early Intervention) program will not have it re-administered.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Change in parental sensitivity | Baseline, Week 10
  Parent sensitivity (warmth, positive regard, respect for child autonomy) will be coded from video-taped parent-child interactions during two play activities. Sensitivity will be coded on a 1 to 7 Likert scale, with higher scores indicating higher sensitivity.

SECONDARY OUTCOMES:
Change in use of higher-level versus lower-level language strategies | Baseline, Week 10
  Parents use of higher level language strategies (open-ended questions, parallel talk, expansion) during video-taped parent-child interactions will be coded. Parent interactions will be transcribed and the number of specific language strategies will recorded.
Change in parental involvement and self-efficacy | Baseline, Week 10
  Parent involved self-efficacy will be measured using the Scale for Parental Involvement and Self-Efficacy (SPISE) for young children with hearing loss. SPISE has a total score ranging from 23 to 161 with the higher score indicating more parent involvement and higher self-efficacy.
Change in Auditory Skills | Baseline, Week 10
  Children's auditory skills will be measured using the Infant-Toddler Meaningful Auditory Integration Scale (IT-MAIS). IT-MAIS has a total score ranging from 0-40 with the higher score indicating better auditory skills.Auditory Integration Scale (IT-MAIS). Higher scores indicated better auditory skills

CONTACTS AND LOCATIONS:
Overall Officials: Ivette Cejas, PhD, Principal Investigator — University of Miami
Locations (1):
- Don Soffer Clinical Research Building, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No